CLINICAL TRIAL: NCT05665426
Title: Effect of Acupuncture or Moxibustion at Acupoints Weizhong (BL40) and Chize (LU5) on the Change in Lumbar Temperature in Healthy People
Brief Title: Infrared Thermography-based Study of the Warming Effect Difference at Waist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Yi Liang, M.D, PhD, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20221101091119441
Record Dates: First submitted 2022-12-14; First posted 2022-12-27 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Health
Keywords: acupuncture; moxibustion; Weizhong; waist
MeSH Terms: interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Intervention Model Description: 2×2 factorial design
Who Masked: Investigator, Outcomes Assessor
Masking Description: The eligible patients will be given a sequential study number by research staff. Subsequently, their basic information will be entered into an internet-based and password-protected clinical research management system (ResMan Research Manager, supported by West China Hospital, Sichuan University, China), which will automatically generate a research code and randomly allocate participants to one of four groups (Acu-BL40 group, Acu-LU5 group, Mox-BL40 group or Mox-LU5 group) at a ratio of 1:1:1:1. Given the nature of the intervention, the participants and acupuncturists will be aware of the assignment. The research assistants responsible for data collection, biostatisticians and data analysis will be masked to study group allocation. Precise documentation of therapy will be recorded in the case report forms (CRFs) in an exclusive computer as well as on paper.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AW group (Other): (1) AW group: acupuncture at Weizhong point,
  Interventions: Other: acupuncture
- AC group (Other): (2) AC group: acupuncture at Chize point,
  Interventions: Other: acupuncture
- MW group (Other): (3) MW group: moxibustion at Weizhong point,
  Interventions: Other: moxibustion
- MC group (Other): (4) MC group: moxibustion at Chize point.
  Interventions: Other: moxibustion

INTERVENTIONS:
Other: acupuncture — Patients allocated to the acupuncture group will be punctured at the pre-specified acupoints. According to the theory of traditional Chinese medicine and clinical experience, we will use the Bilateral Weizhong point (BL 40). Because of the similar anatomy, the Chize point (LU 5) was chosen as a control. Sterile disposable stainless steel acupuncture needles (length: 40 mm, diameter: 0.25 mm; Hwato, Suzhou, China) will be used.
  Arms: AC group; AW group
Other: moxibustion — Moxibustion Participants in the moxibustion group will receive moxibustion treatment via portable Moxibustion (Aikeshu, Bozhou, China); the moxibustion is composed of The inner tube (containing the moxa pillar) and the outer tube. To use, pull out the inner tube and light the moxa pillar, then insert the outer tube and fix the moxibustion on the acupuncture points. Two Moxibustion devices will be sequentially applied at two acupoints Weizhong (BL 40) and Chize (LU 5), for 30 minutes.
  Arms: MC group; MW group

SUMMARY:
Low back pain is a common clinical condition, with up to 84% of adults experiencing varying degrees of low back pain. The most common form of low back pain is non-specific low back pain, which is often treated symptomatically in medicine due to its lack of etiology, which has many side effects. In contrast, acupuncture has the advantage of being practical and free of side effects.

The use of acupuncture points in the lumbar region has a long history of application, as early as the《Huangdi Neijing》thousands of years ago. In the Ming Dynasty, there were summaries of the experience of " Yaobei Weizhong Qiu" (Which means the Weizhong point is closely associated with the waist). Weizhong point's efficacy in lumbar diseases (e.g., lumbar disc herniation, lumbago, sciatica, etc.) is still confirmed. One of the mechanisms is closely related to the improvement of microcirculation, which can be visualized by observing changes in infrared thermal parameters. Acupuncture and moxibustion are the most common therapies at Weizhong point, but there is a lack of research on the differences in efficacy between the two. Therefore, this study aims to collect the temperature parameters of the lumbar region in healthy subjects after acupuncture/moxibustion to estimate the difference in the therapeutic effect on the lumbar region, which can help to reveal the effect differences between acupuncture and moxibustion. As well as to provide scientific evidence to enrich the connotation of the classical theory " Yaobei Weizhong Qiu." the investigators will test the following hypotheses:

1. Hypotheses for main effects of different point selection(LU 5 and BL 40)： H1: There is a significant difference in average temperature change at the waist at 30 minutes between the Weizhong(BL 40) group and the Chize(LU 5) group.

   H0: There is no difference in average temperature change at the waist at 30 minutes between the Weizhong(BL 40) group and the Chize(LU 5) group.
2. Hypotheses for the main effects of different interventions (acupuncture and moxibustion) H1: There is a significant difference in average temperature change at the waist at 30 minutes between the acupuncture group and the moxibustion group.

H0: There is no difference in average temperature change at the waist at 30 minutes between the acupuncture and moxibustion groups.

DETAILED DESCRIPTION:
the investigators will design a 2×2 randomized controlled trial, divided into four groups according to different acupoints (Weizhong and Chize) and different interventions (acupuncture and moxibustion). Patients will be randomized to one of the four treatment arms: (1) AW group: acupuncture at Weizhong point, (2) AC group: acupuncture at Chize point, (3) MW group: moxibustion at Weizhong point, (4) MC group: moxibustion at Chize point. All groups receive the intervention for 30 minutes. This trial will be carried out in the Third Affiliated Hospital of Zhejiang Chinese Medical University. the investigators will measure the average temperature difference of the lumbar region, the average temperature difference of the first lateral line of the Bladder meridian, and the average temperature difference of the second lateral line of the bladder meridian at different time nodes (Pre-intervention, 0, 5, 10, 15, 20, 25, 30 minutes) in all groups.

the investigators used the change of the average temperature (ΔT) in lumbar region from baseline to 30 minutes after intervention as the main effect indicator to estimate the sample size. Sample size calculations are performed to determine the number of participants needed to detect effect sizes. According to previously published results[7, 8] and our preliminary data, the mean and SD of the average temperature difference are μ1 = 0.84 μ2 = 0.34, μ3 = 0.70, and μ4 = 0.20 in the Acu-BL40 group, Acu-LU5 group, Mox-BL40 group and Mox-LU5 group, respectively, with SD σ = 0.26. k represents the number of groups and equals 4 in this trial. Type I error of 5% (α = 0.05) and 80% power (β = 0.20). Estimating a 20% dropout rate during the study, a minimum of 140 total participants is needed to reach the target of 35 participants per group. The investigators will undertake subgroup analysis in BL40 group, according to the pilot study performed previously, although there are about 40% participants can fell the warmth at lumbar region, the ΔT in lumbar region is more significant than others, therefore, the investigators decide not to expand the sample size.

the investigators will recruit 140 eligible participants from Zhejiang Chinese Medical University with age above 18 years. The eligible patients must meet the following inclusion criteria as well as the exclusion criteria. Anticipants will be recruited through an advertisement at the university, and through flyers at several locations of the internet. Interested participants can contact the project leader (PL) through their therapist, by phone or mail. If an applicant meets the study criteria, he or she will be invited to the research.

Temperature detection and measurement Thermal images were obtained using the FLIR E53 camera (FLIR Systems, Inc., Wilsonville, OR, USA). This thermal camera has an infrared resolution of 240×180 pixels and a visible light resolution of 640×480 pixels. The FLIR E53 camera has a scene range temperature range of -20 °C to 650 °C and can detect temperature differences as small as 0.04 °C.

Make the FLIR E53 camera perpendicular to the observing area (pre-marked area and acupoints), from 80 cm. Each participant will be evaluated in a room with a constant temperature of 26°C and 40%-60% humidity. The first photograph will be taken after the participants have rested for 20 min, other photographs will be sequentially taken at 0, 5, 10, 15, 20, 25 and 30 minutes once acupuncture/moxibustion has started and right after the intervention has ended. Heat lamps and other extraneous heat sources are switched off to prevent incorrect measurements.

Thermal images will be analyzed in the FLIR Tools application by two observers. The specific area of interest at the waist as well as the acupoints are predefined and outlined in the normal VGA photograph. The FLIR Tools application allows for calculating the mean temperature in a selected area or line. The mean temperature of certain areas will be compared at different time nodes. The temperature difference between both areas was expressed as ΔT (℃). the investigators will calculate the interobserver reliability by comparing the ΔT value of both researchers.

Interventions. For better observation of temperature changes in the acupoints, KSE36A0R thermometer (Keshun Instrument Co., Ltd., Ningbo, China) will be placed near the acupoint to record the temperature.

This trial will be designed with two interventions of acupuncture and moxibustion, with two acupoints Weizhong (BL 40) and Chize (LU 5) for each intervention. Both acupuncture and moxibustion will be performed by the licensed doctors of traditional Chinese medicine with at least 2 years of experience. Both acupuncture and moxibustion treatment will only consist of 1 session treatment with 30 minutes. Nee dles and moxa will be removed if the patients suffer from any adverse events (AEs).

Adverse Events and Safety All adverse events (AEs) associated with acupuncture and moxibustion would be recorded during the treatment; these AEs include bleeding, hematoma, burns, fainting, serious pain, local infection, etcetera. During the trial, all unexpected adverse events (AEs) will be observed in detail and documented in CRFs. All AEs reported should be analyzed regardless of the investigators' assessments of causality. If serious adverse events happen, the researchers should report to the PL and ethics committee immediately, who will decide on whether the participant needs to withdraw from the study.

Data collection and management Having sought consent, the demographic and baseline characteristic data in CRFs will be completed by a specific RA who is masked to treatment allocation and trained to administer questionnaires in a standardized way. The data consists Gender, age, weight, height, frequency (weekly) of recent low back discomfort, acupuncture/ moxibustion treatment experience and baseline temperature in the waist. Outcome measurement will be measured by the outcome assessors after the intervention. RAs will conduct quality control of data collection and be responsible for data entry. The PL will be responsible for initial data cleaning, identifying, coding, and conversion into the proper format for data analysis. All forms must be dated and signed by the responsible investigator or one of his/her authorized staff members.

Statistical analysis Intention-to-treat (ITT) analysis will be performed regardless of adherence. Microsoft Excel 2016 and IBM SPSS Statistics 23.0 (SPSS Inc., Chicago, IL, United States) will be used in data analysis. Continuous variables (e.g., age, body mass index, temperature, and intensity of warmth) will be represented as the mean ± standard deviation and compared using independent samples t tests. The investigators will use the chi-squared test to analyse the category variables (e.g., gender and sensation of warmth). A P-value alpha < 0.05 (two-sided) will be used to determine statistical significance. After examining the data for normality (Kolmogorov-Smirnov test), the outcome measures will be analysed using ANOVA (assuming normal distribution) or Kruskal-Wallis (non-parametric). Demographic characteristics and other baseline values will be described using descriptive statistics for each group. Subgroup analysis stratified by warming sensation questionnaire (YES or NO). Significant group interactions will be analysed post hoc.

ELIGIBILITY:
Inclusion criteria include:

1. aged 18-60 (either sex);
2. with a BMI of 18.5-23.9 kg/m2;
3. with no history of lower back pain;
4. with normal range of lumbar mobility (including flexion from 75-90 degrees, extension of 30 degrees, lateral bending from 20-35 degrees, and unilateral rotation of 90 degrees);
5. willing to participate in the trial and have signed the informed consent form.

Exclusion criteria:

1. participants with serious heart, liver, kidney, or hematological diseases;
2. women in menses, pregnancy, or lactation;
3. those unable to complete the imaging in prone position (about 40 minutes);
4. those with cognitive impairments;
5. those with a history of lower back trauma or whiplash within a week;
6. those with skin diseases or skin lesions, sensory impairments, scarring, or neoplasms at the test site;
7. those with metal allergies
8. those who have participated in other clinical trials that may affect the results of the study within the last three weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liang, PhD, Principal Investigator — The Third Affiliated Hospital of Zhejiang Chinese Medicial University
Locations (1):
- the Ethics Board of The Third Affiliated Hospital of Zhejiang Chinese Medicinal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng SY, Wang XY, Lin LN, Liu S, Huang XX, Liu YY, Yu XS, Pan W, Fang JQ, Liang Y. Lumbar temperature change after acupuncture or moxibustion at Weizhong (BL40) or Chize (LU5) in healthy adults: A randomized controlled trial. J Integr Med. 2025 Mar;23(2):145-151. doi: 10.1016/j.joim.2025.01.004. Epub 2025 Jan 16. PMID 39863500
- [Derived] Zheng S, Shen Q, Lyu Z, Tian S, Huang X, Liu Y, Yu X, Pan W, Nie N, Liang Y, Fang J. Effect of acupuncture or moxibustion at Acupoints Weizhong (BL40) or Chize (LU5) on the change in lumbar temperature in healthy adults: A study protocol for a randomized controlled trial with a 2 x 2 factorial design. PLoS One. 2023 Oct 30;18(10):e0291536. doi: 10.1371/journal.pone.0291536. eCollection 2023. PMID 37903112

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AW Group | AC Group | MW Group | MC Group
Started | 35 | 35 | 35 | 35
Completed | 35 | 35 | 35 | 35
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AW Group | AC Group | MW Group | MC Group | Total
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (3.6) | 21.86 (2.0) | 23 (3.2) | 22.3 (1.8) | 22.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 27 | 32 | 115
  Male | 6 | 8 | 8 | 3 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 35 | 33 | 34 | 35 | 137
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 3
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline-Mean BMI [Mean (Standard Deviation); unit: kg/m2] | 20.4 (2.4) | 20.2 (2.6) | 20.4 (1.7) | 20.4 (1.7) | 20.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: ΔT at the Waist Between 30 Minutes and the Baseline.
Description: The temperature difference (ΔT)at the waist between 30 minutes and the baseline.
Time Frame: 30 minutes after the intervention has begin
Measure: Mean (Standard Deviation); unit: ℃
Arm/Group | AW Group | AC Group | MW Group | MC Group
Number analyzed (Participants) | 35 | 35 | 35 | 35
℃ | 0.71 (0.67) | 0.42 (0.60) | 0.43 (0.60) | 0.49 (0.65)

2. Secondary Outcome: δT of The Maximum Temperature in the Designated Area of the Waist After 30 Minutes.
Description: The change temperature (δT) of The maximum temperature in the designated area of the waist after 30 minutes.
Time Frame: 30 minutes after the intervention has begin
Measure: Mean (95% Confidence Interval); unit: ℃
Arm/Group | AW Group | AC Group | MW Group | MC Group
Number analyzed (Participants) | 35 | 35 | 35 | 35
℃ | 0.57 [0.37 to 0.77] | 0.41 [0.21 to 0.60] | 0.41 [0.23 to 0.59] | 0.48 [0.31 to 0.66]

3. Secondary Outcome: The Temperature at the Waist Between 5 ,10 ,15 ,20 ,25, 30 Minutes and Baseline.
Description: The temperature between 5 minutes,10 minutes,15 minutes,20 minutes ,25 minutes, 30 minutes and baseline.
Time Frame: 5 minutes,10 minutes,15 minutes,20 minutes,25 minutes , 30 minutes after the intervention has begin
Measure: Mean (Standard Deviation); unit: ℃
Arm/Group | AW Group | AC Group | MW Group | MC Group
Number analyzed (Participants) | 35 | 35 | 35 | 35
℃
  baseline | 34.06 (0.8) | 34.07 (0.88) | 34.16 (0.80) | 33.62 (0.79)
  5 min | 34.32 (0.71) | 34.21 (0.80) | 34.37 (0.72) | 33.80 (0.90)
  10 min | 34.47 (0.69) | 34.34 (0.73) | 34.47 (0.65) | 33.87 (0.73)
  15 min | 34.55 (0.66) | 34.36 (0.70) | 34.53 (0.62) | 33.96 (0.75)
  20 min | 34.59 (0.57) | 34.45 (0.68) | 34.53 (0.61) | 34.02 (0.71)
  25 min | 34.9 (0.62) | 34.50 (0.70) | 34.60 (0.61) | 34.09 (0.71)
  30 min | 34.77 (0.54) | 34.50 (0.70) | 34.59 (0.61) | 34.11 (0.70)

4. Secondary Outcome: ΔT at the Governor Vessel Between 30 Minutes and Baseline
Description: The temperature difference (ΔT) at the Governor Vessel between 30 minutes and baseline
Time Frame: 30 minutes after the intervention has begin
Measure: Mean (95% Confidence Interval); unit: ℃
Arm/Group | AW Group | AC Group | MW Group | MC Group
Number analyzed (Participants) | 35 | 35 | 35 | 35
℃ | 0.49 [0.28 to 0.70] | 0.68 [0.45 to 0.91] | 0.48 [0.22 to 0.74] | 0.41 [0.21 to 0.60]

5. Secondary Outcome: Number of Participants Reporting a Sensation of Warmth in the Lower Back
Description: After completion of the intervention, participants completed a short questionnaire asking whether they experienced a sensation of warmth in the lower back during the intervention (response options: Yes/No). The outcome will be reported as the number and percentage of participants responding "Yes."
Time Frame: Immediately after completion of the intervention session (within 5 minutes of needle withdrawal).
Measure: Count of Participants; unit: Participants
Arm/Group | AW Group | AC Group | MW Group | MC Group
Number analyzed (Participants) | 35 | 35 | 35 | 35
Participants | 12 | 12 | 6 | 11

ADVERSE EVENTS:
Time Frame: Immediately after completion of the intervention session (within 30 minutes of needle withdrawal).
Description: Adverse events were monitored through systematic assessment at each study visit and via participant self-report.
Arm/Group | AW Group | AC Group | MW Group | MC Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 1/35 | 1/35 | 0/35 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2.86% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AW Group (N=35) | AC Group (N=35) | MW Group (N=35) | MC Group (N=35)
Subcutaneous bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05665426/Prot_SAP_000.pdf